CLINICAL TRIAL: NCT02745678
Title: Localized Therapeutics for the Treatment of Gastrointestinal Disorders II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha R Sinha, MD, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB- 34970
Record Dates: First submitted 2016-03-23; First posted 2016-04-20 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Colitis, Ulcerative
Keywords: Enema; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermosensitive gel formulation (Experimental): Thermosensitive gel rectal formulation.
  Interventions: Drug: Thermosensitive gel rectal formulation

INTERVENTIONS:
Drug: Thermosensitive gel rectal formulation

SUMMARY:
The purpose of this study is to investigate a novel thermosensitive topical gel formulation for the treatment of inflammatory bowel disease (IBD), specifically ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign written informed consent.
* Male or non-pregnant and non-lactating females at least 8 years of age.
* Confirmed diagnosis of active, mild to moderate ulcerative proctitis or proctosigmoiditis extending no further than 40cm from the anal verge. Typically, baseline Mayo Disease Activity Index (MMDAI) score between 5 and 10 (indicating mild to moderate disease).

Exclusion Criteria:

* Known infection with Clostridium difficile (C. difficile) and/or other enteric pathogens
* 5-aminosalicylic acid (5-ASA) intolerance
* Current or recent (3 weeks) oral or rectal steroids
* History of thiopurine or Anti-tumor necrosis factor (Anti-TNF) alpha treatment for colitis
* Abnormal creatinine
* Previous small bowel or colonic resection,
* Anal sphincter incompetence,
* Current smokers.
* History or current diagnosis of Crohn's disease or indeterminate colitis.
* History of diverticulitis, collagenous colitis, celiac disease, recurrent pancreatic or known gallbladder disease.
* Unstable significant cardiovascular, endocrine, neurologic or pulmonary disease.
* Hemoglobin levels < 7.5 g/dL.
* History of sclerosing cholangitis, cirrhosis, or hepatic impairment
* Pregnant or at risk of pregnancy.
* Some medications to treat UC are prohibited during participation in the study, including laxatives and anti-diarrhea medications; oral 5-ASA agents and daily fiber supplements are allowed.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of a new formulation in patients with mild-to-moderately-active Ulcerative Colitis using the Mayo Disease Activity Index (MMDAI) | Between 4-6 weeks post-administration
  Using Modified Mayo Score

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No